CLINICAL TRIAL: NCT06545201
Title: RE001 T Cell Injection for the Treatment of KRAS G12V Mutated Solid Tumors, an Open-label Single-center Phase I Clinical Trial
Brief Title: RE001 T Cell Injection for the Treatment of KRAS G12V Mutated Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE00120231204
Record Dates: First submitted 2024-06-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: KRAS G12V; T Cell Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RE001T cell adoptive immunotherapy (Experimental): 3+3 dose increasing design was adopted, and the dose increasing scheme was as follows (deviation 30%): low dose group: 4×109, middle dose group: 8×109, and high dose group: 1.6×1010. If the subjects in the lower dose group continue to benefit clinically after the first T cell infusion treatment, the second T cell infusion treatment can be carried out after the researcher's suggestion and the sponsor's consent. The second infusion can be carried out within 6 months of the disease progression, and the interval between the last infusion and the last infusion is at least 8 weeks.
  Interventions: Biological: RE001 T cell

INTERVENTIONS:
Biological: RE001 T cell — All subjects who met the entry and exit criteria and signed the informed consent form were observed in hospital at the beginning of lymphocyte clearance chemotherapy, with the dosage of cyclophosphamide (600-800mg/m^2/days,-5,-4 days) and fludarabine (25-30mg/m^2/days,-5,-4,-3 days), at least two days after the completion of lymphocyte clearance chemotherapy.

SUMMARY:
At present, there is an urgent need for new drugs for kirsten rat sarcoma viral oncogene (KRAS) mutant tumors in clinic. Preclinical studies support the specificity, safety and anti-tumor activity of RE001. Previous similar studies suggest the feasibility of T cell receptor engineered T cell therapy (TCR-T) treatment, and measures have been taken to ensure the safe administration of RE001 and the close monitoring and management of adverse events. To sum up, RE001 has controllable safety and anti-tumor activity on KRAS mutant solid tumor, which can be preliminarily studied to provide support for clinical research of patients with advanced solid tumor.

DETAILED DESCRIPTION:
This study is a single-center, open, single-arm, dose-increasing, single-dose phase I clinical trial of safety and tolerance. It is planned to recruit 30 patients with advanced malignant solid tumor with KRAS G12V mutation.

In this experiment, 3+3 dose increasing design was adopted, and the dose increasing scheme was as follows (deviation 30%): low dose group: 4×109, middle dose group: 8×109, and high dose group: 1.6×1010. At least 21 days before T cell infusion, peripheral blood mononuclear cell (PBMC) (about 1×10^9) of the subjects were collected by a single blood cell separator. After gene editing, these cells were amplified in vitro and infused into the subjects after reaching the target number. The evaluation period of dose-limited toxicity (DLT) was 28 days after the first administration of each dose group.

The subjects were administered at intervals, and the interval of administration began from the day of TCR-T cell infusion of the previous subject to the day of TCR-T cell infusion of the next subject. The interval between the first three subjects in the same dose group and the next subject (the same group or different groups) is at least 14 days; If one third of the subjects in the dose group have DLT, and three new subjects need to be added, the interval with the next subject (same group or different group) should be at least 21 days.

All the subjects who met the entry and exit criteria and signed the informed consent form were observed in hospital at the beginning of lymphocyte clearance chemotherapy, with the dosage of cyclophosphamide (600-800mg/m^2/days,-5,-4 days) and fludarabine (25-30mg/m^2/days,-5,-4,-3 days), at least two days after the completion of lymphocyte clearance chemotherapy.

During the trial, the subjects can withdraw from the study at any time for any reason, which will not affect the subsequent treatment and care of the subjects by medical staff or medical institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study and sign informed consent;
2. Age ≥18 years old and ≤75 years old;
3. Advanced malignant solid tumors with clear pathological diagnosis;
4. Standard therapies failed or cannot be tolerated or lacks effective treatments;
5. Have at least one measurable lesion;
6. During the trial screening period, the following two indicators must be met (the sponsor is responsible):

   HLA-A* 11:01 positive; Tumor gene testing carries KRAS G12V mutation;
7. ECOG score 0-1 and expected survival time greater than 6 months;
8. Cardiac color ultrasound shows left ventricular ejection fraction ≥50%;
9. Laboratory examination results should meet the following specified indicators:

   White blood cell count ≧ 3.0×109/L;
   1. Absolute neutrophil count ≧ 1.5×109/L (without G-CSF and GM-CSF support, enter at least 14 days before group);
   2. Absolute lymphocyte count ≧ 0.5×109/L;
   3. Platelets (PLT) ≧ 75×109/L (no blood transfusion treatment in the first 14 days);
   4. Hemoglobin ≧ 100g/L (no blood transfusion treatment in the first 14 days);
   5. Prothrombin time international normalized ratio INR ≦ 1.5×upper limit of normal time, unless anticoagulant therapy was received;
   6. Partial prothrombin time (APTT) ≦ 1.5×upper limit of normal time, unless receiving antibiotics coagulation therapy;
   7. Serum creatinine ≦ 1.5mg/dL (or 132.6μmol/L);
   8. Aspartate aminotransferase (AST/SGOT) ≦ 2.5×ULN;
   9. Alanine aminotransferase (ALT/SGPT) ≦ 2.5×ULN;
   10. Total bilirubin (TBIL) ≦ 1.5×ULN;
   11. In patients with liver metastasis, aspartate aminotransferase and alanine aminotransferase need to be ≦ 5×ULN.
10. Women of childbearing age who have not undergone sterilization before menopause must agree to use effective contraception within at least 12 months from the beginning of the study to T cell infusion, and the serum pregnancy test is negative within 14 days before the first treatment;
11. Men who have not undergone sterilization must agree to use effective contraception from the beginning of the study to at least 12 months after T cell infusion;
12. During the entire trial period, you can regularly visit the participating research institutions for relevant testing, evaluation and management.

Exclusion Criteria:

1. Those who have received major surgery, conventional chemotherapy, large-area radiotherapy, immunotherapy or biological therapy anti-tumor treatment within 4 weeks before entering the trial;
2. Previous use of drugs targeting KRAS G12V mutations, including previous participation in cell therapy with similar targets Cellular testing and small molecule inhibitors targeting KRAS G12V mutations, etc.;
3. Allergic reactions are known to occur to any ingredient (such as dimethyl sulfoxide, cyclophosphamide, fludarabine) or structurally similar compounds treated in this trial;
4. Failure to recover from adverse reactions related to previous surgery or treatment to < Grade 2 CTCAEV5.0;
5. Hypertension that remains uncontrolled after combined treatment with 2 drugs or clinically significant (such as active) Cardiovascular and cerebrovascular diseases, such as cerebrovascular accident (within 6 months before signing the informed consent form), myocardial infarction (within 6 months before signing the informed consent form), unstable angina, congestive heart failure classified as class II or above by the New York Heart Association, or severe arrhythmia that cannot be controlled with medication or has a potential impact on study treatment; the electrocardiogram showed obvious abnormality or average QTc interval ≧ 450ms for 3 consecutive times (at least 5 minutes interval);
6. Combined with other serious organic diseases and mental disorders;
7. Suffering from systemic active infections requiring treatment, including but not limited to active tuberculosis, known HIV positive patients or patients with clinically active hepatitis A, B, or C include virus carriers;
8. Have a history of inflammatory bowel disease and autoimmune diseases judged by the researcher to be unsuitable for this study (such as systemic lupus erythematosus, vasculitis, etc.);
9. Those who plan to use the following drugs within 4 weeks before cell therapy and during the study: long-term systemic use steroid hormones, hydroxyurea, immunomodulatory drugs (such as interleukin 2, alpha or gamma interferon, GM-CSF, mTOR inhibitors, cyclosporins, thymosin, etc.);
10. People with brain metastasis:

    1. Symptomatic brain metastasis should be ruled out. Patients with a previous history of symptomatic brain metastasis and stable symptoms after local treatment were enrolled in the group who did not need antiepileptic drugs and steroids at least 14 days before lymphocyte clearance.
    2. Subjects with asymptomatic brain metastasis without tumor-related brain edema, displacement, steroids or antiepileptic drugs can be enrolled.
    3. Subjects with meningitis or meningeal metastasis need to be excluded.
11. People with bleeding or thromboembolism tendency:

    1. Have clinically significant bleeding symptoms or obvious bleeding tendency within 2 weeks before the study;
    2. Have inherited or acquired bleeding and thrombosis tendencies;
    3. A serious arterial/venous thromboembolic event within the past 6 months.
12. Suffering from massive pericardial effusion or symptomatic thoracic or abdominal effusion;
13. Have received live attenuated vaccines within 4 weeks before cell infusion, or plan to receive this type of vaccine during the study;
14. History of organ allogeneic transplantation, allogeneic stem cell transplantation and renal replacement therapy;
15. Uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure;
16. Known alcohol and/or drug abusers;
17. Pregnant or breastfeeding women;
18. Have any coexisting medical conditions or diseases that the researcher determines may impair the conduct of this trial subjects;
19. No legal capacity/restricted capacity;
20. Have previously received any gene or cell therapy products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR). | 24-36 months
  Defined as the proportion of subjects with confirmed CR and PR.

SECONDARY OUTCOMES:
Duration of response (DOR). | 24-36 months
  Defined as the time from cell infusion to disease progression or death in subjects achieving CR or PR.

OTHER OUTCOMES:
Disease control rate (DCR). | 24-36 months
  Defined as the proportion of subjects who achieved CR, PR, and SD after treatment.
Stable disease (DOSD). | 24-36 months
  The definition refers to the period from the start of treatment to the time of evaluation for PD.
Progression-free survival (PFS). | 24-36 months
  Definition refers to the time from the subject's enrollment date (starting treatment date) to the occurrence of PD or death for any reason, whichever occurs first.
Overall survival (OS). | 24-36 months
  Definition refers to the time from the beginning of treatment to death from any cause.
Self-evaluation results of patients. | 24-36 months
  EORTC QLQ-C30 scale was adopted and evaluated according to the scoring manual provided by EORTC.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China